CLINICAL TRIAL: NCT04356521
Title: Lateral Sagittal Versus Costoclavicular Approach for Ultrasound-Guided Infraclavicular Brachial Plexus Block: Comparison of Block Dynamics and Patient Comfort
Brief Title: Lateral Sagittal vs Costoclavicular Approach for Ultrasound-Guided Infraclavicular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Assistant Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC0255
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia, Local; Nerve Block; Brachial Plexus Block
Keywords: Anesthesia, Conduction; Ultrasound; Brachial Plexus Block/methods; Infraclavicular; Costoclavicular approach; Lateral Sagittal approach; Upper Extremity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group LS (Active Comparator): Ultrasound-guided infraclavicular block - lateral sagittal approach (20 ml 0.5% bupivacaine)
  Interventions: Procedure: Lateral Sagittal Approach
- Group CC (Active Comparator): Ultrasound-guided infraclavicular block - costoclavicular approach (20 ml 0.5% bupivacaine)
  Interventions: Procedure: Costoclavicular Approach

INTERVENTIONS:
Procedure: Lateral Sagittal Approach — The US probe will be located medial to the coracoid process in the sagittal plane in the infraclavicular region, and then three cords of the brachial plexus will be viewed. Using the in-plane technique, bupivacaine 0.5% will be administered around the posterior cord (7ml), lateral cord (7ml), and medial cord (6ml).
  Other Names: Infraclavicular Block - Lateral Sagittal Approach
  Arms: Group LS
Procedure: Costoclavicular Approach — The US probe will be placed parallel to the clavicle in the midclavicular area and tilted toward the cephalad and the axillary artery, and three cords will be viewed. A needle will be forwarded from lateral to medial with the in-plane technique, and 20 ml of bupivacaine 0.5% will be administered at the center of the three cords.
  Other Names: Infraclavicular Block - Costoclavicular Approach
  Arms: Group CC

SUMMARY:
An ultrasound-guided infraclavicular block performed with the costoclavicular (CC) approach and the lateral sagittal (LS) approach will be compared in patients scheduled for forearm and hand surgery.

DETAILED DESCRIPTION:
The CC approach is a recently introduced infraclavicular approach that targets three cords (medial, lateral and posterior) located lateral to the axillary artery in the costoclavicular space. Cords in this space are located more superficially than with the classical approach at the lateral infraclavicular fossa and are clustered but maintain a consistent anatomical relationship with each other.

Patients will be divided into two groups:

Group LS: Ultrasound-guided infraclavicular block - lateral sagittal approach (20 ml 0.5% bupivacaine)

Group CC: Ultrasound-guided infraclavicular block - costoclavicular approach (20 ml 0.5% bupivacaine)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 65 years
* Patients scheduled for elective forearm and hand surgeries
* Patients with American Society of Anesthesiologists (ASA) 1-3

Exclusion Criteria:

* Patients not consenting/unwilling to participate
* Age <18 years or >65 years
* Patients with ASA 4
* Obesity (BMI >30 kg/m2)
* Regional anesthesia contraindicated (thrombocytopenia, infection at injection site)
* Severe renal, cardiac, or hepatic disease
* History of hypersensitivity or allergy to local anesthetics
* History of opioid or steroid use for more than 4 weeks
* History of psychiatric disorders
* Analgesic treatment in the last 48 hours preoperatively
* Operations lasting less than 60 minutes and more than 180 minutes
* Patients who converted to general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Performance time of the operator | During the block procedure
  Time elapsed from when the needle enters the skin after an optimal view is obtained on ultrasound until the block needle exits the skin after the procedure is completed.
Duration of start of motor block | 45 minutes after the block procedure
  Time from when a Lovett score of 5 is seen in at least 1 of 3 cords in the patient extremity on which the operation is being performed, following local anesthetic injection.
  Lovett rating scale: 6 = normal muscle strength, 5 = slightly decreased muscle strength, 4 = significantly decreased muscle strength, 3 = slight loss of movement, 2 = significant loss of movement, 1 = near total loss of movement, and 0 = total paralysis.
  Motor block cord myotomes will be evaluated as medial cord (thumb adduction = ulnar nerve), lateral cord (elbow flexion = mucocutaneous nerve), and posterior cord (wrist extension = radial nerve).
Start time of the nervous block | 45 minutes after the block procedure
  Time from the local injection to when a pin-prick test yields no response in at least 1 of 3 cords in the extremity on which the operation is being performed.

SECONDARY OUTCOMES:
Time of sensory block | Postoperative Day 1
  Time when the patient describes pain or when the pin-prick test yields a positive response in the extremity on which the operation is performed.
Time of motor block | Postoperative Day 1
  Time when Lovett score is 2 at any of the 3 dermatomes of the extremity on which the operation is being performed.
  Lovett rating scale 6 = normal muscle strength, 5 = slightly decreased muscle strength, 4 = significantly decreased muscle strength, 3 = slight loss of movement, 2 = significant loss of movement, 1 = near total loss of movement, and 0= total paralysis.
  Motor block cord myotomes will be evaluated as medial cord (thumb adduction=ulnar nerve), lateral cord (elbow flexion= mucocutaneous nerve), and posterior cord (wrist extension=radial nerve).
Patient Satisfaction | Postoperative Day 1
  The discomfort produced by the procedure will be evaluated using the visual rating scale (VRS) at the end of the operation day.
  VRS: 0-100, 0 = no discomfort at all, 100 = excessive discomfort.
Surgeon Satisfaction | Postoperative Day 1
  Surgeon satisfaction will be evaluated at the end of the operation day using the VRS.
  VRS: 0-100, 0 = no discomfort at all, 100 = excessive discomfort.
Number of needle redirections | During the block procedure
  Number of needle redirections until target area is reached: number of attempts to withdraw and redirect the needle without total withdrawal from the skin.
Number of needle attempts | During the block procedure
  Number of needle attempts required until target area is reached: number of withdrawals and redirections of the needle with total withdrawal from the skin.
Number of patients who required a rescue block | 45 minutes after the block procedure
  Patients subjected to an additional rescue block due to positivity in a pin-prick test at a sensorial examination 45 minutes after the block procedure; these patients will be recorded.
Time of first analgesic request | Postoperative Day 1
  Time at which the first analgesic is requested.

CONTACTS AND LOCATIONS:
Overall Officials: BURHAN DOST, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Leurcharusmee P, Elgueta MF, Tiyaprasertkul W, Sotthisopha T, Samerchua A, Gordon A, Aliste J, Finlayson RJ, Tran DQH. A randomized comparison between costoclavicular and paracoracoid ultrasound-guided infraclavicular block for upper limb surgery. Can J Anaesth. 2017 Jun;64(6):617-625. doi: 10.1007/s12630-017-0842-z. Epub 2017 Feb 15. PMID 28205117
- [Background] Songthamwat B, Karmakar MK, Li JW, Samy W, Mok LYH. Ultrasound-Guided Infraclavicular Brachial Plexus Block: Prospective Randomized Comparison of the Lateral Sagittal and Costoclavicular Approach. Reg Anesth Pain Med. 2018 Nov;43(8):825-831. doi: 10.1097/AAP.0000000000000822. PMID 29923950
- [Background] Kavrut Ozturk N, Kavakli AS. Comparison of the coracoid and retroclavicular approaches for ultrasound-guided infraclavicular brachial plexus block. J Anesth. 2017 Aug;31(4):572-578. doi: 10.1007/s00540-017-2359-6. Epub 2017 Apr 18. PMID 28421316
- [Background] Oh C, Noh C, Eom H, Lee S, Park S, Lee S, Shin YS, Ko Y, Chung W, Hong B. Costoclavicular brachial plexus block reduces hemidiaphragmatic paralysis more than supraclavicular brachial plexus block: retrospective, propensity score matched cohort study. Korean J Pain. 2020 Apr 1;33(2):144-152. doi: 10.3344/kjp.2020.33.2.144. PMID 32235015
- [Background] Layera S, Aliste J, Bravo D, Fernandez D, Garcia A, Finlayson RJ, Tran DQ. Single- versus double-injection costoclavicular block: a randomized comparison. Reg Anesth Pain Med. 2020 Mar;45(3):209-213. doi: 10.1136/rapm-2019-101167. Epub 2020 Jan 14. PMID 31941792
- [Background] Mistry T, Balavenkatasubhramanian J, Natarajan V, Kuppusamy E. Ultrasound-guided bilateral costoclavicular brachial plexus blocks for single-stage bilateral upper limb surgeries: Abstain or indulge. J Anaesthesiol Clin Pharmacol. 2019 Oct-Dec;35(4):556-557. doi: 10.4103/joacp.JOACP_222_18. No abstract available. PMID 31920246
- [Background] Monzo E, Hadzic A. Costoclavicular approach to the brachial plexus block: simple or double injection? Reg Anesth Pain Med. 2019 Sep 29:rapm-2019-100852. doi: 10.1136/rapm-2019-100852. Online ahead of print. No abstract available. PMID 31570494
- [Background] Silva GR, Borges DG, Lopes IF, Ruzi RA, Costa PRRM, Mandim BLDS. [Ultrasound-guided costoclavicular block as an alternative for upper limb anesthesia in obese patients]. Braz J Anesthesiol. 2019 Sep-Oct;69(5):510-513. doi: 10.1016/j.bjan.2019.01.004. Epub 2019 Sep 10. PMID 31519300